CLINICAL TRIAL: NCT05688865
Title: Correlation and Clinical Utility of Urinary Biomarker in Membranous Glomerulonephritis
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheuk-Chun SZETO, Professor, Department of Medicine & Therapeutics, Chinese University of Hong Kong
Other Study IDs: CRE-2022.642
Record Dates: First submitted 2023-01-08; First posted 2023-01-18 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Membranous Nephropathy
Keywords: glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis, Membranous; Glomerulonephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urinary cell-free DNA fragments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: urinary markers — urinary marker testing

SUMMARY:
To assess the correlation of these urinary biomarkers with the serum sample and evaluated the clinical utility of using urinary sample in the detection and prognostication of MGN. Fifty patients with newly diagnosed biopsy proven MGN would be recruited and followed up for 1 years. Serum and urinary biomarkers would be collected every 4 months and their antibody titres measured with ELISA assay.

DETAILED DESCRIPTION:
The uses of phospholipase A2 receptor and thrombospondin domain containing 7A antibodies have transformed the management of membranous glomerulonephritis (MGN). However, these are mostly based on serum and the utility of urinary biomarkers are yet to be established.

The aim of this study is to assess the correlation of these urinary biomarkers with the serum sample and evaluated the clinical utility of using urinary sample in the detection and prognostication of MGN. Fifty patients with newly diagnosed biopsy proven MGN would be recruited and followed up for 1 years. Serum and urinary biomarkers would be collected every 4 months and their antibody titres measured with ELISA assay.

The primary outcome would be the correlation of the urinary biomarkers with the corresponding serum markers. The secondary outcome would be the correlation of the urinary biomarkers with clinical parameters such as the slope of eGFR decline, composite renal events such as time to need for renal replacement therapy or renal death and response to treatments.

By establishing the clinical correlation of these urinary biomarkers, the use of such biomarkers would be a more attractive option given its non-invasive nature and conveniences as compared to serum samples.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed biopsy proven primary membranous glomerulonephritis

Exclusion Criteria:

* secondary causes of membranous nephropathy, e.g. lupus nephritis, viral hepatitis B and C and malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to recruit 50 patients with newly diagnosed biopsy proven primary membranous glomerulonephritis. The pathologic diagnosis of membranous nephropathy is made by light microscopy, immunofluorescence including PLA2R/ THSD7A staining and electron microscopy. Secondary causes would be excluded after extensive clinical workup including detailed medical history and patient examination, serological markers of systemic autoimmunity. Essentially, lupus nephritis, viral hepatitis B and C and malignancy would be excluded. The severity of the primary membranous glomerulonephritis is defined according to the KDIGO clinical practice guideline on glomerular diseases.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
serum anti-PLA2R levels | 12 months
rate of renal function decline | 12 months
  eGFR decline

SECONDARY OUTCOMES:
progression to end stage kidney disease | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine & Therapeutics, Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No